CLINICAL TRIAL: NCT03722381
Title: Evaluation of Amlodipine Pharmacokinetics in Patients Receiving Hi Flux Hemodialysis
Status: Withdrawn | Type: Observational
Why Stopped: Study activities were not initiated, and we do not plan to initiate them in the future.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Amy Barton Pai, Amy Pai, PharmD Associate Professor, University of Michigan
Other Study IDs: HUM00143303
Record Dates: First submitted 2018-10-09; First posted 2018-10-26 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Hemodialysis; Pharmacokinetics
MeSH Terms: interventions — Amlodipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Amlodipine Besylate — Pharmacokinetics

SUMMARY:
The current study will evaluate the plasma pharmacokinetics of amlodipine in a cohort of 8 adult volunteers who are receiving regular hemodialysis treatment (HD) 3 days a week for 4 hours each day and have been taking a total daily dose of 5-10 mg of amlodipine besylate for >30 days as part of their usual care. Blood sampling will occur over 13 hours, with frequent sampling during HD and in the 4 hours after termination of HD treatment. The 8 subjects will all receive their prescribed total daily dose of 5-10 mg 5 hours prior to HD treatment. The pre-HD sample will also be sent for pharmacogenomics genotyping. Safety and pharmacodynamic assessments (blood pressure (BP) and heart rate (HR) assessments) will be performed throughout the study. Axiom Precision Medicine Research Array (Affymetrix, Santa Clara, CA) will be used to evaluate genotype of CYP3A4. CYP3A4 phenotype will be evaluated using the ratio of parent drug to metabolite. Non-compartmental analyses will be performed to compare maximum concentrations (Cmax), time to maximum concentration and area under the curve from time 0 to the last measurable sample (AUClast) between the two phases. Compartmental analyses will be performed to construct a model to explain time-dependent changes in amlodipine clearance. Monte Carlo simulations will be performed to compare amlodipine pharmacokinetic profiles on and off HD.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Indwelling tunneled catheter, AVF, AVG that is currently used for hemodialysis
3. Receiving in-center hemodialysis 3 days a week for 3-4.5 hours each treatment
4. Taking a total daily dose of 5-10 mg of amlodipine as prescribed by their physician
5. Hemoglobin ≥ 9.5 g/dL on most recent laboratory assessment prior to study

Exclusion Criteria:

1. Any condition that would not allow for arm BP to be taken
2. Hemoglobin < 9.5 g/dL on most recent lab prior to study
3. Patient is on a CYP3A4 inhibitor (most common in HD population include: amiodarone, clarithromycin, cyclosporine, diltiazem, erythromycin, fluconazole, fluoxetine, fluvoxamine, nefazodone, tamoxifen, verapamil, and grapefruit juice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory in-center hemodialysis patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Use pharmacokinetics to characterize the plasma concentration of amlodipine and its metabolite, 2-([4-(2-chlorophenyl)-3-ethoxycarbonyl-5-methoxycarbonyl-6-methyl- 2-pyridyl]methoxy) acetic acid | Pre-dialysis, during dialysis (30 minutes, 2 hours, end of treatment) and post-dialysis (30 minutes, 2 hours and 4 hours)
  Use pharmacokinetics to characterize the change in plasma concentration of amlodipine and its metabolite, 2-([4-(2-chlorophenyl)-3-ethoxycarbonyl-5-methoxycarbonyl-6-methyl- 2-pyridyl]methoxy) acetic acid during and after HD

SECONDARY OUTCOMES:
Characterize the Non-renal clearance phenotype and genotype | 30 minutes
  Evaluate the non-renal clearance of amlodipine in patients on HD.
Characterize the Post-dialysis Rebound | post-dialysis (30 minutes, 2 hours and 4 hours)
  Simulate change in predicted rebound of metoprolol concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Dialysis, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No